CLINICAL TRIAL: NCT05227053
Title: STOP AF First Post-Approval Study, an Addendum to the Cryo Global Registry
Brief Title: STOP AF First Post-Approval Study
Status: Recruiting | Type: Observational
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: STOP AF First PAS
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Arctic Front™ Cardiac Cryoablation Catheter — Pulmonary vein isolation will be performed with the Arctic Front™ cardiac cryoablation catheter system

SUMMARY:
The STOP AF First PAS is a prospective, global, multi-center, observational trial.

DETAILED DESCRIPTION:
The STOP AF First Post Approval Study (PAS) is a sub-study to the Cryo Global Registry. The STOP AF First PAS is a prospective, global, multi-center, observational trial. The purpose of the study is to describe long-term clinical performance and safety data in the recurrent symptomatic paroxysmal AF population treated with Arctic Front™ and Freezor™ MAX Families of cardiac cryoablation catheters (hereafter referred to as Arctic Front™ Cardiac Cryoablation Catheter System) as an alternative to antiarrhythmic drug therapy as an initial rhythm control strategy. This PAS is a condition of the pre-market approval order (P100010/S110) by the U.S. Food and Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with symptomatic paroxysmal AF
* Subject is ≥ 18 years of age or minimum age as required by local regulations
* Planned pulmonary vein isolation (PVI) procedure using the commercially available Arctic Front™ cardiac cryoablation catheter System.
* Willing to comply with study requirements and give informed consent (defined as legally effective, documented confirmation of a subject's voluntary agreement to participate in this clinical study) or authorization per institution and geographical requirements

Exclusion Criteria:

History of AF treatment with a class I or III antiarrhythmic drug, including sotalol, with the intention to prevent an AF recurrence1

. Subjects under the following conditions may be included in the study:

1. Temporary treatment with a class I or III AAD (treatment at a therapeutic dose for a period of <4 weeks prior to the index PVI procedure)
2. Recent treatment with a class I or III AAD (within 6 months of the index PVI procedure) at a dose below therapeutic threshold according to the AHA/ACC/HRS Guideline for the Management of Patients with Atrial Fibrillation
3. A subject who has received a chemical cardioversion may be included in the study. This includes a chemical cardioversion prior to enrollment and between enrollment and ablation.

   * Subject has had a prior atrial ablation (except for cavo-tricuspid isthmus (CTI) ablation for AFL)
   * Subject is enrolled in a concurrent study that has not been approved for concurrent enrollment by the global study manager
   * Subject with exclusion criteria required by local law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects ≥ 18 years of age (or minimum age as required by local regulations) who have a recommendation for a pulmonary vein ablation with the Arctic Front™ cardiac cryoablation catheter System.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Freedom from Atrial Fibrillation (AF) /Atrial Flutter (AFL) /Atrial Tachycardia (AT) | 36 months
  Estimate the 36-month freedom from Atrial Fibrillation (AF) /atrial flutter (AFL) /Atrial Tachycardia (AT) recurrence using the Arctic Front™ cardiac cryoablation catheter System.
Freedom from Primary Safety Events | 12 months
  Estimate primary safety Adverse Event (AE) rates for cryoablation using the Arctic Front™ cardiac cryoablation catheter System through 12-months.

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun Tarakji, MD, Study Director — Medtronic CAS Chief Medical Officer
Locations (13):
- United States (13):
  - Alaska Heart Institute, Anchorage, Alaska
  - Cardiology Associates of Fairfield County, Stamford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - BayCare Medical Group Cardiology, Clearwater, Florida
  - Heart Rhythm Solutions, Davie, Florida
  - Iowa Heart, West Des Moines, Iowa
  - Our Lady of the Lake, Baton Rouge, Louisiana
  - Southcoast Health System, North Dartmouth, Massachusetts
  - Henry Ford Heart & Vascular, Detroit, Michigan
  - The Lindner Research Center, Cincinnati, Ohio
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - University of Tennessee Methodist Physicians, Memphis, Tennessee
  - Texas Health Research and Education Institute, Dallas, Texas